CLINICAL TRIAL: NCT02611557
Title: Imaging Noninvasively With Functional-MRI for Onset, Response and Management of Lymphatic Impairment
Brief Title: Lymphedema Progression Screening Using MRI
Acronym: INFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Manus Donahue, Associate Professor of Radiology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Donahue_Lymphedema
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Lymphedema; Breast Cancer
Keywords: MRI; lymphedema; manual lymphatic drainage
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manual lymphatic drainage therapy (Other): Patients will undergo a 50 min manual lymphatic drainage (MLD) therapy session by a certified lymphedema therapist. MLD therapy is performed routinely for standard of care in these patients and consists of light massage to facilitate lymphatic fluid mobility.
  Interventions: Procedure: Manual lymphatic drainage therapy

INTERVENTIONS:
Procedure: Manual lymphatic drainage therapy — Patients will undergo a 50 min manual lymphatic drainage (MLD) therapy session by a certified lymphedema therapist. MLD therapy is performed routinely for standard of care in these patients and consists of light massage to facilitate lymphatic fluid mobility.

SUMMARY:
This study will apply novel, noninvasive structural and functional magnetic resonance imaging (MRI) methods to patients with mild and moderate breast cancer-related lymphedema (BCRL) for the first time to test fundamental hypotheses about relationships between lymphatic compromise and imaging biomarkers that may portend disease progression and individualized therapy response.

DETAILED DESCRIPTION:
Lymphedema is a chronic, debilitating disease caused by lymphatic flow obstruction. Breast cancer-related lymphedema (BCRL) secondary to mastectomy and/or radiation therapy is a growing health concern, with a reported incidence as high as 94% in breast cancer survivors. Behavioral adjustments and aggressive therapeutic management can reduce long-term impairment and optimize quality of life. However, there is currently no standard clinical procedure for identifying patients at greatest BCRL risk and fundamental gaps exist in even our basic knowledge of how the lymphatic system responds to node dissection and subsequent therapy. Specialized imaging methods have demonstrated that reduced lymphatic flow velocity and lymphatic contractility impairment may signify greater BCRL risk, however these approaches frequently require radioactive tracers or exogenous contrast agents which alter the physiological environment and are primarily available only in specialized centers. As such, these methods are simply impractical for routine BCRL monitoring in humans or for reporting clinical trial endpoints.

Recent work has demonstrated that spin labeling, a popular and noninvasive MRI method for measuring perfusion, can be adapted to measure lymphatic fluid flow to axillary lymph nodes. Furthermore chemical exchange saturation transfer (CEST) MRI, a popular method for measuring protein content and pH changes in brain, breast, and liver, can be translated to the lymphatic system to assess sensitive changes in interstitial protein accumulation, a hallmark of lymphedema progression. Recent work has provided motivation for these techniques by demonstrating, using commercially available equipment, that consistent changes in lymphatic properties are detectable in vivo under (i) conditions of cuff-induced lymph flow manipulation, and (ii) in affected vs. unaffected arms of BCRL patients. Here, these methods will be implemented in sequence with standard clinical and MRI measures of lymph structure to expand our understanding of lymph physiology in different stages of BCRL and in response to therapy.

Hypothesis (1). Axillary lymph nodes and vessels, velocity of lymphatic fluid, and interstitial protein accumulation can be visualized in a reproducible manner using noninvasive MRI approaches that are frequently used to measure analogous metrics in brain, breast, and liver.

Aim (1). Turbo-spin-echo, spin labeling, and CEST MRI will be applied to assess lymph collector volume, lymphatic flow velocity, and interstitial protein accumulation, respectively, together for the first time in healthy female volunteers. Intraclass and Spearman's rank correlation coefficients will be calculated to understand the reproducibility and age-dependence of these parameters in uncompromised lymphatic systems.

Hypothesis (2). (2a) The MRI protocol applied in Aim (1) can be used to detect (i) increases in interstitial protein accumulation and (ii) reductions in lymphatic velocity in patients with mild and moderate BCRL, and (2b) these functional metrics will be more variable than limb volume measurements in patients in early BCRL disease stages and following common manual lymphatic drainage (MLD) therapy, thereby demonstrating the utility of these imaging biomarkers for identifying lymphatic dysfunction and monitoring therapy response.

Aim (2). The Aim (1) protocol will be applied to patients in preclinical (Stage 0), mild (Stage I), and moderate (Stage II) BCRL together with volumetric limb measurements before and after MLD therapy. A Wilcoxon rank-sum test will be used to assess differences in parameters between patient volunteers in different BCRL stages as well as pre- and post-MLD therapy. These data will provide an exemplar for how the novel, internal imaging measurements of lymphatic function vary with disease severity and therapy administration.

Hypothesis (3). In preclinical BCRL patients (Stage 0), reduced lymphatic velocity and increased interstitial protein accumulation correlates with elevated two-year BCRL progression risk.

Aim (3). Stage 0 BCRL patients will undergo an identical MRI protocol as outlined in Aim (1) and follow-up disability metrics will be recorded up to two years post-therapy. A multi-parametric analysis will be used to test correlations between the hypothesized imaging biomarkers and BCRL progression, thereby demonstrating to what extent acute MRI may be used to stratify risk in patients at high risk for BCRL.

This work will for the first time translate a noninvasive, multi-modal MRI protocol, which has demonstrated clinical potential in brain, liver, and breast applications, to the human lymphatic system to better characterize lymphatic dysfunction, therapy response, and BCRL risk in the growing breast cancer survivor population.

ELIGIBILITY:
Inclusion Criteria:

* sex=female
* age=40-70 yrs
* clinical diagnosis of lymphedema secondary to breast cancer treatment (including node dissection, radiation therapy, and/or sentinel node biopsy).

Exclusion Criteria:

* Contraindication to MRI
* Bilateral axillary lymph node removal
* Primary lymphedema. Individuals on tyrosine kinase inhibitors or calcium channel blockers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Lymphedema progression | 2 years
  Progression to more advanced stage of lymphedema. Stage 0 to Stage 1 criteria: ≥ 2 cm difference in arm circumference between involved and uninvolved arms. Fibrosis: none or minimal; Pitting: pits on pressure; Elevation: reduces edema; Skin: no change. Stage I to II progression criteria: Stage I circumference criteria with Fibrosis: moderate; Pitting: may be present; Elevation: does not fully reduce edema (minimal to no reduction); Skin: no change. All progression will be determined using the Perometer by a certified lymphedema therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Manus J Donahue, PhD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Result] Donahue MJ, Donahue PC, Rane S, Thompson CR, Strother MK, Scott AO, Smith SA. Assessment of lymphatic impairment and interstitial protein accumulation in patients with breast cancer treatment-related lymphedema using CEST MRI. Magn Reson Med. 2016 Jan;75(1):345-55. doi: 10.1002/mrm.25649. Epub 2015 Mar 7. PMID 25752499
- [Result] Rane S, Donahue PM, Towse T, Ridner S, Chappell M, Jordi J, Gore J, Donahue MJ. Clinical feasibility of noninvasive visualization of lymphatic flow with principles of spin labeling MR imaging: implications for lymphedema assessment. Radiology. 2013 Dec;269(3):893-902. doi: 10.1148/radiol.13120145. Epub 2013 Oct 28. PMID 23864103
- [Result] Donahue PM, Crescenzi R, Scott AO, Braxton V, Desai A, Smith SA, Jordi J, Meszoely IM, Grau AM, Kauffmann RM, Sweeting RS, Spotanski K, Ridner SH, Donahue MJ. Bilateral Changes in Deep Tissue Environment After Manual Lymphatic Drainage in Patients with Breast Cancer Treatment-Related Lymphedema. Lymphat Res Biol. 2017 Mar;15(1):45-56. doi: 10.1089/lrb.2016.0020. PMID 28323572
- [Result] Crescenzi R, Donahue PMC, Hartley KG, Desai AA, Scott AO, Braxton V, Mahany H, Lants SK, Donahue MJ. Lymphedema evaluation using noninvasive 3T MR lymphangiography. J Magn Reson Imaging. 2017 Nov;46(5):1349-1360. doi: 10.1002/jmri.25670. Epub 2017 Feb 28. PMID 28245075
- [Derived] Crescenzi R, Donahue PMC, Garza M, Lee CA, Patel NJ, Gonzalez V, Jones RS, Donahue MJ. Elevated magnetic resonance imaging measures of adipose tissue deposition in women with breast cancer treatment-related lymphedema. Breast Cancer Res Treat. 2022 Jan;191(1):115-124. doi: 10.1007/s10549-021-06419-w. Epub 2021 Oct 23. PMID 34687412